CLINICAL TRIAL: NCT04327713
Title: Systematic Review and Meta-analysis of Randomized Controlled Trials of the Effect of Fish Oil Supplementation on Cardiovascular Outcomes in Diabetes
Brief Title: Meta-analysis of Fish Oil Supplementation and Cardiovascular Outcomes in Diabetes
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Collaborators: Diabetes and Nutrition Study Group (DNSG) of the European Association for the Study of Diabetes (EASD) (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government); Diabetes Canada (Other)
Responsible Party: Principal Investigator, John Sievenpiper, Associate Professor, University of Toronto
Other Study IDs: DNSG-Fish oil
Record Dates: First submitted 2020-03-28; First posted 2020-03-31 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Type2 Diabetes; Heart Failure; Myocardial Infarction; Stroke; Arrhythmia; Cardiovascular Diseases
Keywords: fish oil supplementation; Cardiovascular disease; stroke; myocardial infarction; diabetes; coronary heart disease; systematic review; meta-analysis
MeSH Terms: conditions — Heart Failure; Myocardial Infarction; Stroke; Arrhythmias, Cardiac; Cardiovascular Diseases; Diabetes Mellitus; Coronary Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- fish oil supplementation: fish oil supplementation, usually capsules with a defined content of EPA and DHA
  dosage and duration of intervention differ between the included studies of our meta-analysis
  Interventions: Dietary Supplement: fish oil supplement
- placebo supplementation: placebo supplementation, usually capsules with a defined content of non-fish oil or other components
  content, dosage and duration of intervention differ between the included studies of our meta-analysis
  Interventions: Dietary Supplement: fish oil supplement

INTERVENTIONS:
Dietary Supplement: fish oil supplement — daily fish oil supplement vs. placebo

SUMMARY:
Fish oil contains a large amount of long-chain omega-3 polyunsaturated fatty acids, which are considered an important component of a healthy diet. As many patients do not eat fish, supplementation with fish oil is a common strategy to provide sufficient amounts of these particular fatty acids in daily life. Fish oil supplementation has been investigated for decades for its cardio-protective effects and its ability to lower serum triglycerides. People with diabetes mellitus have an increased risk for cardiovascular events and show alterations in lipids with high triglycerides. Whether there is a benefit of fish oil supplementation in this high risk group remains unclear with major international diabetes associations recommending against the use of fish oil supplements. The European Association for the Study of Diabetes (EASD) has not made any recommendations about the use of fish oils in people with diabetes since 2004. To inform the update of the EASD clinical practice guidelines for nutrition therapy, the Diabetes and Nutrition Study Group (DNSG) of the EASD has commissioned the proposed systematic review and meta-analysis of randomized controlled trials of the effect of fish oil supplementation on cardiovascular outcomes in people with diabetes and use the Grading of Recommendations Assessment, Development and Evaluation (GRADE) approach to assess the certainty of the evidence.

DETAILED DESCRIPTION:
Background: Cardiovascular disease (CVD) accounts for a large proportion of annual deaths around the world. In both the general population as well as in high-risk subgroups, achieving a healthy diet is one approach to lower the risk for CVD. Fish oil supplements have been widely investigated for cardiovascular indications, showing consistent reductions in triglycerides with variable effects on other intermediate risk factors (glycemia, blood pressure, inflammation) which have not translated into reductions in patient-important clinical outcomes. Recent systematic reviews and meta-analyses of the available randomized trials have failed to show a meaningful cardiovascular benefit of fish oil supplementation. It is unclear whether this lack of benefit holds across all groups, especially groups with a high triglyceride phenotype and at high cardiovascular risk such as those with diabetes. No systematic review and meta-analysis has specifically synthesized the evidence of the effect of fish oil supplementation on cardiovascular outcomes in people with diabetes. On the basis of several recent large cardiovascular outcomes trials in people with diabetes or that included subgroups of people with diabetes, the 2019 American Diabetes Association and 2018 Diabetes Canada clinical practice guidelines recommended against the use of fish oil supplementation for cardiovascular risk reduction in people with diabetes. The European Association for the Study of Diabetes (EASD) have made a similar recommendation but have not updated their clinical practice guidelines since 2004. To inform the update of the EASD clinical practice guidelines for nutrition therapy, the Diabetes and Nutrition Study Group (DNSG) of the EASD has commissioned a series of evidence syntheses. The proposed systematic review and meta-analysis of randomized controlled trials will assess the effect of fish oil supplementation on cardiovascular outcomes in people with diabetes and use the Grading of Recommendations Assessment, Development and Evaluation (GRADE) approach to assess the certainty of the evidence.

Need for proposed research: There is an urgent need for a synthesis of the evidence of the effect of fish oil supplementation on cardiovascular outcomes in people with diabetes to inform the update of the EASD clinical practice guidelines for nutrition therapy. High quality systematic reviews and meta-analyses of randomized controlled trials with assessment of the certainty of the evidence using GRADE provide the strongest form of evidence synthesis to support clinical practice guidelines and public health policy development.

Objective: To inform the update of the European Association for the Study of Diabetes (EASD) clinical practice guidelines for nutrition therapy, the investigators will conduct a systematic review and meta-analysis of randomized controlled trials of the effect of fish oil supplementation on cardiovascular outcomes in people with diabetes and use the GRADE approach to assess the certainty of the evidence.

Design: The planning and conduct of the proposed meta-analyses will follow the Cochrane handbook for systematic reviews of interventions. The reporting will follow the Preferred Reporting Items for Systematic Reviews and Meta-Analyses (PRISMA) guidelines.

Data sources: MEDLINE, EMBASE, and The Cochrane Central Register of Controlled Trials databases will be searched using appropriate search terms supplemented by hand searches of references of included studies.

Study selection: Randomized controlled trials conducted in humans with a follow-up duration ≥ 52 weeks investigating the effect of fish oil supplementation compared to placebo on cardiovascular outcomes will be included. Eligible studies will be conducted in people with diabetes or contain data from a subgroup of people with diabetes. Studies that are not randomized, have a shorter duration (<52 weeks), use multi-modal interventions that do not allow for the isolation of the effect of fish oil supplementation, provide fish oil in the form of a prescription pharmaceutical drug (e.g. icopsant ethyl), lack a suitable control group/comparator, are not conducted in people with diabetes, and/or do not report viable cardiovascular outcomes data will be excluded.

Data extraction: Two investigators will independently extract relevant data and assess risk of bias using the Cochrane Risk of Bias tool Version 2. Events and total participants in intervention group and control groups will be extracted. When avaialble, risk ratios, odds ratios and hazard ratios for clinical outcomes will be extracted or derived from clinical event data across exposure to either fish oil supplementation or placebo. All disagreements will be resolved by consensus. Corresponding authors of relevant publications will be asked for additional data if needed.

Outcomes: The primary outcome will be total CVD incidence. Secondary outcomes will be major adverse cardiovascular events (MACE), CVD mortality, all-cause mortality, coronary heart disease (CHD) incidence, CHD mortality, MI incidence, stroke incidence, and arrhythmia.

Data synthesis: Risk ratios of clinical outcomes using total events and number of people in intervention and control groups will be calculated for each RCT. Reported relative ratio measures will be used for studies not reporting raw numbers and hazard ratio and odds ratios will be considered equivalent to risk ratios.

Data will be pooled using the Mantel-Haenszel method with random effects models. Results will be reported as pooled risk ratios with 95% confidence intervals (95% CI). Heterogeneity will be assessed by the Cochrane Q statistic and quantified by the I2 statistic with I2>50% and P(Q) <0.1 considered evidence of substantial heterogeneity.

If there are ≥10 trials, a priori subgroup analyses will be undertaken to explore sources of heterogeneity including sex, age, type of diabetes (type 1 or type 2 diabetes), prevention type (primary, secondary), intervention type (supplements, supplemented foods, dietary advice), comparator, study design, follow-up duration,baseline glycemic control, risk of bias, funding source. Significant unexplained heterogeneity will be investigated by additional post hoc subgroup analyses. Meta-regression analyses will assess the significance of subgroups analyses.

Sensitivity analysis will be performed by removing one study at a time. A study will be considered influential if it changes the direction or significance of effect and/or heterogeneity.

If there are ≥10 trials, publication bias will be assessed by the inspection of funnel plots and using Begg's and Egger's tests. If publication bias is suspected, we will attempt to adjust for funnel plot asymmetry by imputing the missing study data using the Duval and Tweedie trim and fill method.

Evidence Assessment: The certainty of the evidence for each outcome will be assessed using the Grading of Recommendations Assessment, Development and Evaluation (GRADE) approach.

Knowledge translation plan: The results will be disseminated through talks or posters at regional, national, and international scientific meetings and publication in high impact factor journals. We will target public health and scientific communities interested in nutrition, cardiovascular diseases and diabetes. Their feedback will be incorporated in order to improve the public health message and to define key areas for future research.

Applicant/Co-applicant: Decision Makers will network among opinion leaders to increase awareness and participate directly as committee members in the development of future guidelines.

Significance: The proposed project will aid in knowledge translation related to the role of fish oil supplementation in the prevention of cardiovascular diseases in the high-risk group of T2DM patients, strengthening the evidence-base for guidelines and improving health outcomes by educating healthcare providers and patients, stimulating industry innovation, and guiding future research design.

ELIGIBILITY:
Inclusion Criteria:

* Randomized controlled trials
* Participants with diabetes
* Follow-up duration ≥ 52 weeks
* Intervention involves fish oil supplementation using supplements, supplemented foods, or dietary advice
* Control group
* Ascertainment of at least one cardiovascular outcome

Exclusion Criteria:

* Non-randomized studies
* Participants without diabetes
* Follow-up duration <52 weeks
* Multi-modal interventions
* Interventions of fish oils in the form of a prescription pharmaceutical drug (e.g. icosapent ethyl)
* Lack of a suitable control group (e.g. fish oil containing comparator)
* No viable cardiovascular outcome data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with type 2 diabetes mellitus
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2020-03-28 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Total cardiovascular disease (CVD) incidence | at least 1 year
  Risk ratio of fatal and non-fatal CVD events

SECONDARY OUTCOMES:
Major adverse cardiovascular events (MACE) | at least 1 year
  Risk ratio of MACE
CVD mortality | at least 1 year
  Risk ratio of fatal CVD events
All-cause mortality | at least 1 year
  Risk ratio of all-cause mortality
Coronary heart disease (CHD) incidence | at least 1 year
  Risk ratio of fatal and non-fatal CHD events
Coronary heart disease (CHD) mortality | at least 1 year
  Risk ratio of fatal CHD events
Myocardial infarction (MI) incidence | at least 1 year
  Risk ratio of fatal and non-fatal MI events
Stroke incidence | at least 1 year
  Risk ratio of fatal and non-fatal stroke events
Arrhythmia incidence | at least 1 year
  Risk ratio of fatal and non-fatal arrhythmia events

CONTACTS AND LOCATIONS:
Overall Officials: John L Sievenpiper, MD,PhD,FRCPC, Principal Investigator — University of Toronto
Locations (1):
- Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
We don't have access to individual participant data, as we are conducting a systematic review and meta-analysis.